CLINICAL TRIAL: NCT05147012
Title: Intraoperative Hypotension Predicted by Observation of Mean Arterial Pressure : a Retrospective Cohort Preliminary Study
Brief Title: Intraoperative Hypotension Predicted by Mean Arterial Pressure
Acronym: HYPPOPOPAM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: HYPPOPOPAM_2020
Record Dates: First submitted 2020-06-12; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2020-06

CONDITIONS: Wedge Resection; Lobectomy by Video-thoracoscopies
Keywords: wedge resection; lobectomy; video-thoracoscopies
MeSH Terms: interventions — Routinely Collected Health Data

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control group
- focus group
  Interventions: Other: Data collected

INTERVENTIONS:
Other: Data collected — The variable of the characteristic of the patients (i.e.: age, sex, hypertension, diabetes, atrial fibrillation, coronary arteries diseases, body mass index (BMI), surgery, medications) were retrieved from the anesthesia consultation file (Easily, Hospices Civiles de Lyon, France).
  We retrieved the mean arterial pressure from our local anesthesia software for each patient ( Diane®, Bow medical, Amiens France). We also performed an automatic extraction of data from our anesthesia software (Diane, Bow Medical, France) with a rate of 1 value / minute for some continuous arterial pressure.
  All data was extracted from our institutional database and collected by a physician who was not involved in the care of the study patients.
  Groups: focus group

SUMMARY:
During general anesthesia, intraoperative hypotension (IOH) is associated with increased morbidity and mortality. Mean arterial pressure (MAP) < 65mmHg is the most common definition of hypotension. In order to reduce IOH, a complex method using machine learning called hypotensive prediction index (HPI) was shown to be superior to changes in MAP (ΔMAP) to predict hypotension (MAP between 65 and 75 excluded). Linear extrapolation of MAP (LepMAP) is also very simple and could be a better approach than ΔMAP. The main objective of the present study was to investigate whether LepMAP could predict IOH during anesthesia 1, 2 or 5 minutes before.

Hypothesis : the area under the ROC curves (ROC Area Under Curves) at 1, 2 and 5 minutes of LepMAP would be superior to ΔMAP

ELIGIBILITY:
Inclusion Criteria:

* All lobectomy including for another study (VATOFA study) with continuous invasive blood pressure monitoring per arterial line
* All pancreaticoduodenectomy or hepatectomy including for another study (CARBODAV study) with continuous invasive blood pressure monitoring per arterial line
* age 18 or over

Exclusion Criteria:

* complex hemodynamic cases (heart, lung and liver transplantation)
* using extracorporeal membrane oxygenation.
* Patient who object to take part of the study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all gender minimum age : 18 years old Healthy volunteers are not accepted
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
AUC ROC of LepMAP | Only during perioperative period
  The primary outcome measure is the AUC ROC of LepMAP 1, 2 and 5 minute before hypotension to predict hypotension defined as a mean arterial pressure less tha 65 mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Intensive Care, Louis Pradel University Hospital, Bron, France

IPD SHARING:
Plan to Share IPD: No